CLINICAL TRIAL: NCT02850081
Title: Statin Neuroprotection and Carotid Endarterectomy: Safety, Feasibility and Outcomes
Acronym: STANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AAAM2407
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Carotid Artery Stenosis; Strokes
Keywords: Carotid endarterectomy; CEA; stroke; asymptomatic stenosis
MeSH Terms: conditions — Carotid Stenosis; Stroke | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Observational - Maximal Dose - ARM 1 (No Intervention): Patients on a pre-existing maximal dose of either Simvastatin (40mg) with/without currently taking amlodipine (Norvasc) and those on Simvastatin 20mg while currently on amlodipine; Atorvastatin (80mg), or Rosuvastatin (20mg) regimen will be observed for ~2 weeks before their CEA.
- Less Than Maximal Dose - ARM 2 (Experimental): Patients on a pre-existing statin regimen at a lower dose (less than maximal) of Simvastatin <40mg without amlodipine and <20mg with amlodipine; Atorvastatin (<80mg) or Rosuvastatin (<20mg) will be randomized to maintain their current dose plus placebo or be increased to the maximal dose of their current statin for ~2 weeks before their CEA.
  Interventions: Drug: Statin; Other: Placebo
- Statin Naive - ARM 3 (Experimental): Patients on no pre-existing statin regimen will be randomized to Atorvastatin 10 mg or Atorvastatin 80 mg for ~2 weeks before their CEA
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Statin — Standard of care treatment (one of four):
  * Simvastatin (to 40mg without amlodipine)
  * Simvastatin (to 20 mg if currently on amlodipine)
  * Atorvastatin (to 80mg)
  * Rosuvastatin (to 20mg)
  Other Names: Pre-existing statin regimen
  Arms: Less Than Maximal Dose - ARM 2
Drug: Atorvastatin — A lipid-lowering agent and for prevention of events associated with cardiovascular disease.
  10 mg or 80 mg capsules
  Other Names: Lipitor
  Arms: Statin Naive - ARM 3
Other: Placebo — A placebo pill will be used for patients that are to maintain their current dose of statins prior to their CEA.
  Other Names: Sugar pill
  Arms: Less Than Maximal Dose - ARM 2

SUMMARY:
The investigators hypothesize that pre-operative statin use is neuroprotective at maximal doses. The goals are to determine the safety, feasibility, and efficacy of maximizing statin doses for two weeks (12-18 days) prior to CEA using change in performance on a battery neuropsychometric tests as outcome measure. Study will recruit patients based on their preexisting statin regimen.

The investigators hypothesize that in asymptomatic CEA patients: 1) Pre-operative statin use is neuroprotective against early cognitive dysfunction (eCD) and lowers the risk of early mortality. 2) Maximal doses may be essential in achieving optimal neuroprotection against eCD.

DETAILED DESCRIPTION:
Carotid endarterectomy (CEA) is a common surgery performed to reduce the risk of stroke in patients with carotid artery narrowing. Statins, a class of drugs usually used to lower blood cholesterol, may protect the brain after surgery. Specific statins have been shown to protect the brain after surgery when compared to others. eCD affects about 25% of patients undergoing CEA and about 15% of undergoing asymptomatic CEA. It is associated with marked elevations in tissue markers of cerebral injury and is associated with earlier post-CEA mortality. This clinically significant, but subtle, cerebral injury is 10 times more common than stroke and its mechanism appears to be similarly related to regional hypoperfusion and ischemia. It is imperative to determine in a prospective randomized trial whether alteration/increase of preoperative statin regimens leads to improved neurologic outcome and an even lower incidence of stroke and possibly greater survival.

In order to optimally design and conduct such a trial it is critical to: 1) explore the safety and feasibility of altering statin regimen acutely (approximately 2 weeks) before CEA, and 2) clearly establish the neuroprotective outcome of an acute alteration in statin regimen. This would promote a better understanding of statin neuroprotection in humans and determine the statin treatment that affords the most neuroprotection in patients undergoing one of the most commonly performed procedures in the US.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age.
2. Patient is currently on atorvastatin or simvastatin or rosuvastatin or statin naïve (no statins in the last 30 days).
3. The patient has unilateral or bilateral carotid artery stenosis that is considered severe (carotid artery diameter reduction ≥ 70%) as defined by:

   1. Peak systolic velocity of at least 230 cm/s plus at least one of these:
   2. End diastolic velocity ≥ 100 cm/s OR
   3. CTA showing ≥ 70% stenosis OR
   4. MRA showing ≥ 70% stenosis
4. This stenosis has not caused any stroke, transient cerebral ischemia, or other relevant neurological symptoms in the past.
5. The patient's attending doctor(s) (PMD, cardiologist, vascular/neurosurgeon) AND the patient have decided to proceed with a CEA to treat the patient's severe carotid stenosis.
6. The patient has no known circumstance or condition likely to preclude 1 year follow-up or adherence to the study protocol.
7. The patient is independent in their Activities of Daily Living at baseline.
8. Patient has the ability to provide informed consent.

Exclusion Criteria:

1. Patient has underlying disease other than atherosclerosis (i.e. autoimmune disease, known active malignancy).
2. Patient has documented dementia or screens out based on abnormal Baseline MoCA (≤25) and AD8 (≥2).
3. Patient's life expectancy is < 12 months.
4. Patient has advanced renal failure (serum creatinine > 2.5 mg/dL)
5. Patient has evidence of severe congestive heart failure or has history of end-stage cardiovascular disease (e.g. CHF NYHA Class III or IV or unstable angina).
6. Patient has history of intolerance or allergic reaction to any statins (myotoxicity, hepatic dysfunction, rash, etc.)
7. Patient has received an investigational drug within 30 days.
8. Patient is pregnant or lactating.
9. Patient is currently taking any of the following which have been shown to interact with atorvastatin and/or simvastatin and/or rosuvastatin (as per current drug package inserts):

   * Cyclosporine;
   * HIV Protease Inhibitors/Antivirals (e.g. rotanavir or plus rotanavir, tipranavir, lopinavir, boceprevir, saquinovir, darunavir, fosamprenavir, nelfinavir, efavirenz/tenofobir, atazanavir, simeprevir);
   * Hep C Protease Inhibitor/Antivirals (e.g. telapravir);
   * Antibiotics (i.e. cobicistat-containing products like Tybost, rifampin/rifampicin, clarithromycin, telithromycin, erythromycin);
   * Anti-fungals (i.e. itraconazole, ketoconazole, posaconazole, voriconazole, fluconazole); *Gemfibrozil; Other Fenofibrates (e.g. Tricor, fibric acid);
   * Niacin > 1g/day or statins in combination with niacin (e.g. Vytorin, Simcor);
   * Colchicine;
   * Danazol;
   * Calcium Channel Blockers: Diltiazem, Varapamil;
   * Dronedarone;
   * Amiodarone;
   * Digoxin;
   * Ranolazine;
   * Nefazodone;
   * Warfarin/Coumadin;
   * Lomitapide;
   * Grapefruit juice > 1.2 liters/day (40.5 ounces/day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Prevalence of eCD | 30 Days: 1) Pre-op vs. Post-CEA Day 1 (12-25 hrs post-op) and 2) Pre-op vs. Post-CEA Day 30
  Neurocognitive assessments ≥2SD worse than reference group in two or more cognitive domains or (b) ≥1.5SD worse than the reference group in all cognitive domains.

SECONDARY OUTCOMES:
Prevalence of early mortality | 1 year
  Data will be collected by follow up phone call

CONTACTS AND LOCATIONS:
Overall Officials: Edward S Connolly, MD, FACS, Principal Investigator — Columbia University Medical Center/New York Presbyterian; Eric Heyer, MD, Ph.D., Study Director — Columbia University
Locations (7):
- United States (7):
  - Valley Hospital, Ridgewood, New Jersey
  - Albany Medical College/The Vascular Group at Albany, Albany, New York
  - State University of New York at Buffalo, Buffalo, New York
  - New York University School of Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cornell University Medical College (Weill), New York, New York

IPD SHARING:
Plan to Share IPD: No